CLINICAL TRIAL: NCT02957266
Title: Improvement of Locally Advanced Cervical Cancer Radiotherapy Efficacy by Use of Volumetric Arc Therapy, Individualized Polyradiosensitization and Interstitial Brachytherapy
Brief Title: Cervical Cancer Radiotherapy by Use of VMAT, Individualized Polyradiosensitization and Interstitial Brachytherapy
Acronym: CERVIPIB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The National Center of Oncology, Azerbaijan (Other Government)
Responsible Party: Principal Investigator, Kamal Akbarov, Radiation Oncologist, PhD, The National Center of Oncology, Azerbaijan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOM-0001
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; interstitial brachytherapy; gemcitabine; volumetric arc therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Cisplatin; Gemcitabine; Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classical treatment (Active Comparator): Classical concurrent cisplatin based chemoradiotherapy of cervical cancer. PIK3CA, KRAS, BRAF and RRM1 mutations rates.
  Interventions: Radiation: Volumetric Arc Radiotherapy; Drug: Cisplatin; Genetic: PIK3CA; Genetic: KRAS; Genetic: BRAF; Genetic: RRM1
- GemInterBraVMAT (Experimental): Concurrent chemoradiotherapy of cervical cancer patients treated by VMAT (volumetric arc radiotherapy) based external beam radiotherapy, polyradiosensitization by cisplatin and gemcitabine and interstitial brachytherapy.
  PIK3CA, KRAS, BRAF and RRM1 mutations rates.
  Interventions: Radiation: Volumetric Arc Radiotherapy; Radiation: Interstitial brachytherapy; Drug: Cisplatin; Drug: Gemcitabine; Genetic: PIK3CA; Genetic: KRAS; Genetic: BRAF; Genetic: RRM1

INTERVENTIONS:
Radiation: Volumetric Arc Radiotherapy — Volumetric Arc Radiotherapy
Radiation: Interstitial brachytherapy — Interstitial High Dose Rate Brachytherapy
  Arms: GemInterBraVMAT
Drug: Cisplatin — Weekly Cisplatin
  Other Names: CDDP
Drug: Gemcitabine — Weekly Gemcitabine
  Other Names: Gemcitabine Hydrochloride
  Arms: GemInterBraVMAT
Genetic: PIK3CA — PIK3CA mutations rate
Genetic: KRAS — KRAS mutations rate
Genetic: BRAF — BRAF mutations rate
Genetic: RRM1 — RRM1 mutations rate

SUMMARY:
The purpose of this study is to define an effectiveness of concurrent chemoradiotherapy of cervical cancer patients treated by VMAT (volumetric arc therapy) based external beam radiotherapy, polyradiosensitization by cisplatin and gemcitabine and interstitial brachytherapy.

DETAILED DESCRIPTION:
Now cisplatin based concurrent chemoradiotherapy for cervical cancer is a standard treatment modality. But we consider that the treatment results could be improved by several ways: 1. use of VMAT (volumetric arc therapy) based external beam radiotherapy could decrease toxicity by reducing of unnecessarily irradiated tissue volumes; 2. in addition to cisplatin gemcitabine could enhance tumor cell damaging effect of radiation; 3. interstitial brachytherapy could provide higher radiation dose boost to high risk tumor volume while sparing surrounding organs at risk.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed primary invasive carcinoma of the uterine cervix Previously untreated disease Any cell type Stage IB2, IIA, IIB, IIIA, IIIB, or IVA Para-aortic lymph nodes negative by radiologic evaluation or by biopsy if CT scan is suspicious for adenopathy No known metastases to scalene nodes or other organs outside the radiotherapy field Study enrollment within 8 weeks of diagnosis Performance status - GOG 0-2 Absolute neutrophil count at least 1,500/mm^3 Platelet count at least 100,000/mm^3 Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Creatinine less than 2.0 mg/dL No renal abnormalities (e.g., pelvic kidney, horseshoe kidney, or renal transplantation) that would require modification of radiotherapy fields No bilateral ureteral obstruction allowed unless treated with stent or nephrostomy tube Not pregnant Fertile patients must use effective contraception No septicemia or severe infection No circumstance that would preclude study completion or follow-up No other malignancy within the past 5 years except nonmelanoma skin cancer No prior cytotoxic chemotherapy No prior pelvic or abdominal radiotherapy No prior therapy for this malignancy

Exclusion Criteria:

Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events.(Note: Serum Pregnancy tests must be obtained in women of child bearing potential). Sexually active females may not participate unless they have agreed to use an effective contraceptive method (such as abstinence, diaphragm, condom, or intrauterine device) to prevent pregnancy for the duration of the study.

Growth factor(s): Growth factors that support platelet or white cell number or function must not have been administered within the past 28 days.

Erythropoietic drug(s): Erythropoietin or related hormones must not have been administered within the past 28 days.

Infection: Patients who have an uncontrolled infection. Evidence of distant metastases Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years.

Prior systemic chemotherapy within the last three years. Prior radiotherapy to the pelvis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Relapse Rate (local and/or distant) and Number of Deaths Due to Any Cause | 4 years

SECONDARY OUTCOMES:
Number of Participants With Progressive Disease | 4 years
Incidence of acute toxicity | Up to 30 days after completion of radiation therapy
Incidence of late toxicity | Up to 2 years after completion of radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Akbarov, PhD, Principal Investigator — National Center of Oncology
Locations (1):
- National Center of Oncology, Baku, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: No